CLINICAL TRIAL: NCT01358760
Title: Dehydroepiandrosterone (DHEA) Against Vaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-234
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Vaginal Atrophy
Keywords: Vulvar/vaginal atrophy; Atrophic Vaginitis; Dehydroepiandrosterone; DHEA; Prasterone; Vaginorm; Menopause; Intrarosa
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 0.25% DHEA (Experimental)
  Interventions: Drug: DHEA
- 0.5% DHEA (Experimental)
  Interventions: Drug: DHEA

INTERVENTIONS:
Drug: Placebo — Placebo vaginal suppository
  Arms: Placebo
Drug: DHEA — Vaginal suppository containing 0.25% (3.25 mg) DHEA
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.25% DHEA
Drug: DHEA — Vaginal suppository containing 0.5% (6.5 mg) DHEA
  Other Names: Prasterone, Dehydroepiandrosterone
  Arms: 0.5% DHEA

SUMMARY:
The purpose of this Phase III trial is to evaluate the efficacy of intravaginal dehydroepiandrosterone (DHEA) in postmenopausal women with vaginal atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (non-hysterectomized or hysterectomized)
* Women between 40 and 75 years of age
* Willing to participate in the study and sign an informed consent
* Women who have self-identified symptom(s) of vaginal atrophy
* For non-hysterectomized women, willing to have endometrial biopsy at baseline and end of study

Exclusion Criteria:

* Undiagnosed abnormal genital bleeding
* Hypertension equal to or above 140/90 mm Hg
* The administration of any investigational drug within 30 days of screening visit
* Endometrial hyperplasia, cancer or endometrial histology showing proliferative, secretory or menstrual type characteristics at histologic evaluation of endometrial biopsy performed at screening

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Archer, MD, Principal Investigator — Clinical Research Center, Eastern Virginia Medical School, Norfolk, VA
Locations (42):
- United States (32):
  - EndoCeutics site # 39, Montgomery, Alabama
  - EndoCeutics site # 14, Tucson, Arizona
  - EndoCeutics site # 65, Little Rock, Arkansas
  - EndoCeutics site # 21, Sacramento, California
  - EndoCeutics site # 30, San Diego, California
  - EndoCeutics site # 36, Denver, Colorado
  - EndoCeutics site # 52, Denver, Colorado
  - EndoCeutics site # 66, Danbury, Connecticut
  - EndoCeutics site # 42, Milford, Connecticut
  - EndoCeutics site # 57, West Hartford, Connecticut
  - EndoCeutics site # 61, Newark, Delaware
  - EndoCeutics site # 26, Jacksonville, Florida
  - EndoCeutics site # 60, Lake Worth, Florida
  - EndoCeutics site # 54, North Miami, Florida
  - EndoCeutics site # 56, Pinellas Park, Florida
  - EndoCeutics site # 23, Sandy Springs, Georgia
  - EndoCeutics site # 10, Meridian, Idaho
  - EndoCeutics site # 55, Wichita, Kansas
  - EndoCeutics site # 27, Baltimore, Maryland
  - EndoCeutics site # 24, Omaha, Nebraska
  - EndoCeutics site # 50, Neptune City, New Jersey
  - EndoCeutics site # 33, Beachwood, Ohio
  - EndoCeutics site # 05, Cleveland, Ohio
  - EndoCeutics site # 47, Cleveland, Ohio
  - EndoCeutics site # 15, Columbus, Ohio
  - EndoCeutics site # 62, Providence, Rhode Island
  - EndoCeutics site # 64, Jackson, Tennessee
  - EndoCeutics site # 63, Memphis, Tennessee
  - EndoCeutics site # 53, San Antonio, Texas
  - EndoCeutics site # 51, Sandy City, Utah
  - EndoCeutics site # 09, West Jordan, Utah
  - EndoCeutics site # 03, Norfolk, Virginia
- Canada (10):
  - EndoCeutics site # 13, Calgary, Alberta
  - EndoCeutics site # 06, Bathurst, New Brunswick
  - EndoCeutics site # 59, Toronto, Ontario
  - EndoCeutics site # 04, Drummondville, Quebec
  - EndoCeutics site # 12, Montreal, Quebec
  - EndoCeutics site # 02, Québec, Quebec
  - EndoCeutics site # 01, Québec, Quebec
  - EndoCeutics site # 18, Saint Romuald, Quebec
  - EndoCeutics site # 08, Shawinigan, Quebec
  - EndoCeutics site # 11, Sherbrooke, Quebec

REFERENCES:
- [Result] Bouchard C, Labrie F, Archer DF, Portman DJ, Koltun W, Elfassi E, Grainger DA, Ayotte N, Cooper TA, Martens M, Waldbaum AS, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Decreased efficacy of twice-weekly intravaginal dehydroepiandrosterone on vulvovaginal atrophy. Climacteric. 2015;18(4):590-607. doi: 10.3109/13697137.2014.992012. Epub 2015 Mar 3. PMID 25511551
- [Result] Portman DJ, Labrie F, Archer DF, Bouchard C, Cusan L, Girard G, Ayotte N, Koltun W, Blouin F, Young D, Wade A, Martel C, Dube R; other participating members of VVA Prasterone Group. Lack of effect of intravaginal dehydroepiandrosterone (DHEA, prasterone) on the endometrium in postmenopausal women. Menopause. 2015 Dec;22(12):1289-95. doi: 10.1097/GME.0000000000000470. PMID 25968836

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 897 subjects were screened at 42 medical/research sites located in the US (32 centers) and Canada (10 centers) and 450 subjects were randomized. The first subject first visit was on 21-JUN-2011 and the last subject last visit was on 12-APR-2012.
Groups:
- Placebo: Placebo: Placebo vaginal suppository; daily dosing with one suppository for 2 weeks followed by twice weekly dosing for 10 weeks.
- 0.25% DHEA: DHEA (prasterone): Vaginal suppository containing 0.25% (3.25 mg) DHEA; daily dosing with one suppository for 2 weeks followed by twice weekly dosing for 10 weeks.
- 0.50% DHEA: DHEA (prasterone): Vaginal suppository containing 0.50% (6.5 mg) DHEA; daily dosing with one suppository for 2 weeks followed by twice weekly dosing for 10 weeks.
Period: Overall Study
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Started | 152 | 148 | 150
Safety Population | 150 | 143 | 148
ITT Population | 139 | 134 | 134
Completed | 130 | 128 | 125
Not Completed | 22 | 20 | 25
Not completed — Adverse Event | 3 | 4 | 3
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Entry criteria not met/Non-compliance | 12 | 12 | 16

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population corresponds to the Safety Population which includes all subjects who received any amount of DHEA (prasterone) or placebo, and who have any safety information available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA | Total
Number analyzed (Participants) | 150 | 143 | 148 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.59 (6.47) | 58.41 (6.02) | 58.33 (6.16) | 58.11 (6.22)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 150 | 143 | 148 | 441
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White caucasian | 135 | 132 | 131 | 398
  Black or African American | 12 | 9 | 13 | 34
  Asian | 1 | 1 | 1 | 3
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Other | 1 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of parabasal cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses were performed primarily on the Intent to Treat (ITT) population defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria.
Measure: Mean (Standard Error); unit: percentage of parabasal cells
Groups:
- 0.50% DHEA: DHEA (prasterone): Vaginal suppository containing 0.5% (6.5 mg) DHEA; daily dosing with one suppository for 2 weeks followed by twice weekly dosing for 10 weeks.
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
percentage of parabasal cells
  Baseline | 60.66 (3.40) | 56.74 (3.69) | 59.54 (3.41)
  Week 12 | 62.22 (3.49) | 39.23 (3.15) | 33.02 (3.09)
  Change from Baseline to Week 12 | 1.56 (1.98) | -17.51 (2.74) | -26.52 (2.94)

2. Primary Outcome: Change From Baseline to Week 12 in Percentage of Superficial Cells in the Maturation Index of the Vaginal Smear
Description: The percentage of superficial cells was determined from the vaginal smears collected during the study. A 100-cell count was performed by a central laboratory to classify cells as parabasal (P) (including basal), intermediate (I), and superficial (S) squamous cell types. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of superficial cells
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
percentage of superficial cells
  Baseline | 0.97 (0.13) | 1.12 (0.13) | 0.93 (0.11)
  Week 12 | 1.80 (0.29) | 3.43 (0.34) | 3.58 (0.41)
  Change from Baseline to Week 12 | 0.83 (0.26) | 2.31 (0.32) | 2.66 (0.41)

3. Primary Outcome: Change From Baseline to Week 12 in Vaginal pH
Description: A pH strip fixed on an Ayre spatula (or equivalent) was applied directly to the lateral wall of the vagina. The change in color of the pH indicator strip was compared to the color chart for pH evaluation. The corresponding pH value (with one decimal) was recorded. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pH units
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
pH units
  Baseline | 6.34 (0.05) | 6.27 (0.06) | 6.29 (0.06)
  Week 12 | 6.06 (0.08) | 5.69 (0.09) | 5.67 (0.08)
  Change from Baseline to Week 12 | -0.28 (0.06) | -0.58 (0.07) | -0.62 (0.07)

4. Primary Outcome: Change From Baseline to Week 12 in Severity of the Most Bothersome Symptom of Vaginal Dryness
Description: The severity of vaginal dryness was evaluated by a questionnaire filled out by women. The severity of dryness recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
Severity score
  Baseline | 2.38 (0.04) | 2.37 (0.04) | 2.35 (0.04)
  Week 12 | 1.27 (0.07) | 1.10 (0.07) | 1.13 (0.08)
  Change from Baseline to Week 12 | -1.12 (0.08) | -1.28 (0.08) | -1.22 (0.08)

5. Secondary Outcome: Change From Baseline to Week 12 in Severity of Dyspareunia
Description: The severity of dyspareunia was evaluated by a questionnaire filled out by women. The severity of dyspareunia recorded as none, mild, moderate or severe was analyzed using the score values of 0, 1, 2 or 3, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: Efficacy analyses on dyspareunia were performed on a subgroup of the Intent to Treat (ITT) population (defined as all subjects who have received at least one dose of study drug with a baseline (Day 1) evaluation meeting the study entry criteria) who had self-identified moderate to severe dyspareunia at Baseline.
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 99 | 93 | 100
Severity score
  Baseline | 2.56 (0.05) | 2.58 (0.05) | 2.60 (0.05)
  Week 12 | 1.78 (0.11) | 1.48 (0.12) | 1.54 (0.10)
  Change from Baseline to Week 12 | -0.78 (0.10) | -1.10 (0.12) | -1.06 (0.10)

6. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Secretions
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal secretions (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy were analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
Severity score
  Baseline | 2.71 (0.05) | 2.55 (0.06) | 2.55 (0.06)
  Week 12 | 2.33 (0.06) | 2.07 (0.08) | 2.07 (0.06)
  Change from Baseline to Week 12 | -0.38 (0.05) | -0.48 (0.08) | -0.48 (0.07)

7. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Integrity
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal epithelial integrity (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
Severity score
  Baseline | 2.32 (0.07) | 2.19 (0.07) | 2.19 (0.08)
  Week 12 | 1.94 (0.07) | 1.74 (0.07) | 1.69 (0.07)
  Change from Baseline to Week 12 | -0.38 (0.06) | -0.46 (0.07) | -0.50 (0.08)

8. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Epithelial Surface Thickness
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal epithelial surface thickness (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
Severity score
  Baseline | 2.78 (0.06) | 2.66 (0.06) | 2.72 (0.06)
  Week 12 | 2.40 (0.07) | 2.25 (0.07) | 2.16 (0.06)
  Change from Baseline to Week 12 | -0.38 (0.06) | -0.40 (0.07) | -0.56 (0.07)

9. Secondary Outcome: Change From Baseline to Week 12 in Severity of Vaginal Atrophy as Evaluated From Vaginal Color
Description: To evaluate the aspect of the mucosa and the local tolerance to prasterone ovules, the vaginal color (one of the four main signs of vaginal atrophy) evaluated by the physician/gynecologist as corresponding to none, mild, moderate, or severe atrophy was analyzed using the score values of 1, 2, 3 and 4, respectively. Data obtained at Baseline and Week 12 as well as the change from Baseline to Week 12 are presented.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Severity score
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Number analyzed (Participants) | 139 | 134 | 134
Severity score
  Baseline | 2.66 (0.05) | 2.60 (0.06) | 2.65 (0.06)
  Week 12 | 2.31 (0.07) | 2.16 (0.07) | 2.12 (0.06)
  Change from Baseline to Week 12 | -0.35 (0.06) | -0.45 (0.07) | -0.53 (0.07)

ADVERSE EVENTS:
Time Frame: From Baseline to Week 12 (+ 30-day follow-up period after last dose)
Arm/Group | Placebo | 0.25% DHEA | 0.50% DHEA
Serious Adverse Events (participants affected / at risk) | 5/150 | 1/143 | 1/148
Other Adverse Events (participants affected / at risk) | 19/150 | 17/143 | 23/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | 0.25% DHEA (N=143) | 0.50% DHEA (N=148)
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | 0.25% DHEA (N=143) | 0.50% DHEA (N=148)
Nasopharyngitis (Infections and infestations) | 10 | 7 | 9
Urinary tract infection (Infections and infestations) | 9 | 10 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall provide to the SPONSOR 30 days prior to submission all documents for publication, presentation, etc that report any trial results. The SPONSOR shall have editorial rights on documents and the right to review/comment with regard to (1) proprietary information, (2) accuracy of the information, (3) correctness of the scientific evaluation/conclusions and (4) to ensure that the information is fairly balanced and in compliance with regulations.